CLINICAL TRIAL: NCT06813274
Title: Multicenter, Double Blind, Randomized, Placebo-controlled Trial to Exploring the Role of Eye-Brain Multimodal Imaging in Diagnosing and Treating Neurovascular Coupling Impairment in Diabetes Mellitus
Brief Title: Multicenter RCT of Eye-Brain Imaging in Diabetes Neurovascular Coupling
Acronym: TCM-MMI
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hejiang Ye (Other)
Responsible Party: Sponsor-Investigator, Hejiang Ye, Professor, Chengdu University of Traditional Chinese Medicine
Organization: Chengdu University of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023ZD001
Record Dates: First submitted 2025-01-26; First posted 2025-02-06 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus; Diabetic Retinopathy; Cognitive Impairment; Neurovascular Coupling
Keywords: Eye-Brain Multimodal Imaging; Neurovascular Coupling Impairment; Diabetes Mellitus; Diabetic retinopathy; Diabetic Cognitive Impairment; Traditional Chinese Medicine
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Retinopathy; Cognitive Dysfunction | interventions — mecobalamin

STUDY DESIGN:
Intervention Model Description: This study adopts a block randomization technique to allocate participants into groups, maintaining a 1:1 ratio between the experimental and control arms.
Who Masked: Participant, Investigator
Masking Description: The randomization sequence is crafted by statistical experts uninvolved in the trial's execution, utilizing SAS9.4 software with a predefined seed and an appropriately chosen block length. To ensure consistency, a third-party manufacturer is contracted to produce both the experimental drug and placebo, adhering to uniform labeling and packaging standards. Subsequently, a pharmacist independent of the trial's operational team blinds the medications in accordance with the established randomization sequence. The investigators dispense the drugs sequentially, adhering to the assigned drug numbers and the chronological order of patient enrollment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants assigned to the experimental group will receive hypoglycemic treatment, accompanied by the administration of Tangshen'an Granules, Ginkgo Leaf Tablets, and Mecobalamin Capsules.
  Interventions: Drug: hypoglycemic treatment; Drug: Tangshen'an Granules; Drug: Ginkgo Leaf Tablets; Drug: Mecobalamin Tablets
- Control Group (Placebo Comparator): Participants assigned to the control group will receive hypoglycemic treatment, accompanied by placebo, Ginkgo Leaf Tablets, and Mecobalamin Tablets.
  Interventions: Drug: hypoglycemic treatment; Drug: Ginkgo Leaf Tablets; Drug: Mecobalamin Tablets; Drug: placebo

INTERVENTIONS:
Drug: hypoglycemic treatment — The diabetes management adheres to the "The 2025 Guidelines for Standards of Diabetes Care" issued by the American Diabetes Association (ADA).
Drug: Tangshen'an Granules — Tangshen'an Granules comprises a meticulously blended mix of Astragalus, Prepared Rehmannia Root, Dodder Seed, Kudzu Root, Millettia Speciosa Champ, Salviae Miltiorrhizae Radix et Rhizoma, Poria Cocos, and Polygala Tenuifolia. Tangshen'an Granules is administered at a dosage of 9g, dissolved in boiling water, and taken three times daily.
  Arms: Intervention Group
Drug: Ginkgo Leaf Tablets — The primary active ingredients of Ginkgo Leaf Tablets are ginkgo flavonoid glycosides and terpene lactones. The prescribed oral dosage is one tablet each time, administered three times a day.
Drug: Mecobalamin Tablets — Mecobalamin Tablets primarily contain mecobalamin, which is a coenzyme-active form of vitamin B12. The prescribed oral dosage is 0.5mg, administered three times a day.
Drug: placebo — The placebo contains 10% of the active ingredients in Tangshen'an Granules, formulated by controlling the concentration to mimic Tangshen'an Granules. The placebo is administered at a dosage of 9g, dissolved in boiling water, and taken three times daily.
  Arms: Control Group

SUMMARY:
This study intends to take the critical pathological mechanism of diabetic neurovascular coupling injury (NCI) as the starting point and utilize multi-modal imaging (MMI) technology of the eyes and brain as a means to conduct in-depth, integrated, and interdisciplinary research with Traditional Chinese Medicine (TCM) syndrome studies. The aim is to establish diagnostic and therapeutic standards for diabetic NCI, based on Eye-Brain Multimodal Imaging technology, providing objective and quantitative evidence for early disease diagnosis and therapeutic effect evaluation. Simultaneously, investigators will conduct multicenter, randomized, placebo-controlled, double-blind clinical trials to systematically investigate the clinical efficacy and safety of Tangshen'an Granule in preventing and treating diabetic NCI. By obtaining high-quality evidence-based data on TCM, this study aims to enhance the level of prevention and treatment with TCM and clinical service capabilities, thereby providing new ideas and directions for research.

DETAILED DESCRIPTION:
Diabetes mellitus(DM) is a prevalent condition that often leads to neurovascular coupling impairment (NCI), which has been shown to be intimately associated with diabetic retinopathy and cognitive decline. Given the critical need for early diagnosis and effective treatment, eye-brain multimodal imaging(MMI) technology has emerged as a promising tool in this field. This study focuses on establishing a comprehensive and standardized approach for diagnosing and treating diabetic NCI through the utilization of eye-brain MMI technology accompanied by assessing the effectiveness and potential therapeutic benefits of the traditional Chinese medicine compound, Tangshen'an Granule, in the management of diabetic NCI.

A pool of standard diagnostic and therapeutic entries for diabetic NCI syndromes using eye-brain MMI technology is planned to be established through database retrieval and refined by expert questionnaire surveys to formulate the relevant standards. A multicenter, randomized, double-blind, placebo-controlled clinical evaluation study of Tangshen'an Granules in treating diabetic NCI (kidney deficiency and blood stasis syndrome) patients from specific hospitals will be conducted. Diagnostic criteria involve diabetes diagnosis and specific requirements of multiple eye-brain imaging and cognitive assessment tools. Eligibility criteria include inclusion and exclusion conditions. Randomization and blinding are properly implemented. The intervention includes basic therapy with different drug administrations in the experimental and control groups. The trial lasts 24 weeks. Primary outcomes are evaluated by various eye-brain imaging and cognitive assessment means. Secondary outcomes involve TCM symptom scores, glycemic indicators, and quality of life questionnaire. Safety indicators are monitored. Data is analyzed using Intent-To-Treat (ITT) analysis.

The study protocol has been approved by the Ethics Committee of the Hospital of Chengdu University of Traditional Chinese Medicine(ethical approval number:2023KL-056). Informed consent is planned to be obtained from all participants. The study results will be reported in academic meetings and peer-reviewed journals to promote the development of diagnostic and treatment standards for diabetic NCI.

ELIGIBILITY:
Inclusion Criteria:

* Participants who comply with the diagnostic criteria for DM according to the World Health Organization in 1999.

  * Participants who fulfill the diagnostic criteria for diabetic NCI.

    ③ Participants who diagnosed with the syndrome of kidney deficiency and blood stasis according to TCM syndrome differentiation.

    ④ Participants who have a glycated hemoglobin(HbA1c) level of ≤9%.

    ⑤ Participants who are aged between 18 and 70 years inclusive, with no gender preference.

    ⑥Participants who sign informed consent form.

Exclusion Criteria:

* Participants exhibiting retinopathy induced by alternative etiological factors (including retinal vein occlusion, age-related macular degeneration(AMD), alongside cognitive impairments stemming from endocrine-metabolic disturbances, sleep disorders.

  * Participants suffering from acute diabetic complications (such as diabetic ketoacidosis, hyperosmolar hyperglycemic state).

    * Participants with significant dysfunction in the heart, liver, kidney, or autoimmune disorders.

      ④Participants unable to cooperate due to mental health issues, intellectual disabilities, or similar conditions that impede their participation in the trial.

      ⑤Participants who are allergic to the intervention used in this study.

      ⑥Participants who have engaged in other trials within the past three months or are currently enrolled in another study.

      ⑦Female participants who are in the process of trying to conceive, are pregnant, or are lactating.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Retinal Nerve Fiber Layer Thickness (RNFL) | From the date of randomization until the end of the 24-week intervention period
  The measurement of Retinal Nerve Fiber Layer Thickness (RNFL) is crucial in ophthalmology. Its main parameter is RNFL thickness, which represents the overall average thickness across the entire measured retinal area and is a fundamental metric for initial assessment with a decrease often linked to optic nerve damage.The measurement is often obtained using optical coherence tomography (OCT), a non-invasive imaging technique that delivers high-resolution, cross-sectional images of the retinal layers.
Foveal Avascular Zone (FAZ) | From the date of randomization until the end of the 24-week intervention period
  Foveal Avascular Zone (FAZ) is a crucial parameter in retinal imaging, particularly for evaluating macular vascular integrity and diagnosing retinal vascular diseases, such as diabetic retinopathy. The key parameter is the FAZ area, which provides a detailed morphological and functional assessment of the foveal microvasculature. This measurement is commonly obtained using optical coherence tomography angiography (OCTA), which offers high-resolution, depth-resolved visualization of the retinal vasculature without the need for dye injection.
Visual Evoked Potential (VEP) | From the date of randomization until the end of the 24-week intervention period
  Visual Evoked Potential (VEP) is a neurophysiological technique used to assess the functional integrity of the visual pathway, from the retina to the visual cortex, by measuring the electrical activity generated in response to visual stimuli. Its main parameter is the latency of the P100 wave, which represents the time delay (in milliseconds) between the presentation of a visual stimulus and the peak of the positive waveform occurring around 100 milliseconds post-stimulus. VEP measurement is typically conducted using an electroencephalogram system equipped with specialized software for stimulus presentation and signal analysis, making it an essential tool for evaluating visual pathway integrity, diagnosing neurological disorders, and monitoring disease progression or treatment efficacy.
Gray matter volume (GMV) | From the date of randomization until the end of the 24-week intervention period
  Gray matter volume (GMV) is a pivotal aspect in neuroimaging research, particularly focusing on the structural properties of the brain. A primary parameter in GMV measurement is the absolute volume, which quantifies the volume occupied by neuronal cell bodies, dendrites, and synapses within specific brain regions. This parameter offers crucial insights into brain development, aging, and the pathophysiology of neurological and psychiatric disorders. The GMV is commonly measured by magnetic resonance imaging (MRI) scanners, specifically high-field strength MRI systems that provide superior spatial resolution and contrast.
Montreal Cognitive Assessment（MoCA）score | From the date of randomization until the end of the 24-week intervention period
  The Montreal Cognitive Assessment (MoCA) score is a widely used cognitive screening tool designed to detect mild cognitive impairment and early stages of dementia. It assesses multiple cognitive domains, including attention, executive functions, memory, language, visuospatial abilities, abstraction, calculation, and orientation. The MOCA scale will be downloaded from the official website (https://www.mocatest.org).The test consists of 30 items, with a maximum score of 30 points, and typically takes 10-15 minutes to administer. A score of 26 or above is generally considered normal, while scores below 26 may indicate cognitive impairment.The MoCA is administered by a trained clinician or researcher who scores the participant's performance based on standardized criteria, providing a comprehensive assessment of cognitive function.
Mini - Mental State Examination（MMSE）score | From the date of randomization until the end of the 24-week intervention period
  The Mini-Mental State Examination (MMSE) score is a widely utilized cognitive screening instrument designed to assess cognitive impairment. It evaluates multiple cognitive domains, including orientation, memory, attention, language, and visuospatial abilities, through a series of questions and tasks. The MMSE will be downloaded from the official website at https://www.parinc.com.The MMSE, administered by a trained investigator, consists of 30 items, with a maximum score of 30 points, and typically takes 5-10 minutes to test. A score of below 24 often indicates cognitive impairment.

SECONDARY OUTCOMES:
Symptom scores in traditional Chinese medicine | From the date of randomization until the end of the 24-week intervention period
  Symptom scores in Traditional Chinese Medicine (TCM) are a systematic approach to quantifying and evaluating clinical manifestations based on TCM theory. These scores, administered by a trained investigator, typically assess a range of symptoms, including but not limited to fatigue, pain, digestive issues, sleep disturbances, emotional states, and specific organ-related dysfunctions, through structured questionnaires or clinical observation. The degree can be scored from mild to severe.
Glucose metabolism indicators:Hemoglobin A1c (HbA1c) | From the date of randomization until the end of the 24-week intervention period
  Hemoglobin A1c (HbA1c) is a critical biomarker used to assess long-term glycemic control in individuals with diabetes, reflecting the average blood glucose levels over the preceding 2-3 months. The measurement of HbA1c include high-performance liquid chromatography (HPLC), immunoassay, and affinity chromatography, each offering high precision and accuracy.
Glucose metabolism indicators:Fasting blood glucose | From the date of randomization until the end of the 24-week intervention period
  Fasting Blood Glucose (FBG) is a fundamental test used to measure blood sugar levels after an individual has fasted for at least 8 hours. It is a key diagnostic tool for assessing glucose metabolism and identifying conditions such as diabetes mellitus, prediabetes, and insulin resistance.The measurement is performed using enzymatic methods, such as glucose oxidase or hexokinase assays, which provide high specificity and accuracy.
Quality of Life Scale (SF-36) | From the date of randomization until the end of the 24-week intervention period
  The SF-36 is a widely utilized questionnaire that measures health-related quality of life including physical functioning, bodily pain, general health perceptions, vitality, social functioning and mental health. It employs a standardized set of questions with weighted response options, enabling the quantification of an individual's health status thus serving as a valuable tool in clinical research, healthcare evaluation, and policy-making.

OTHER OUTCOMES:
Blood Routine Test：White Blood Cell Count (WBC) | From the date of randomization until the end of the 24-week intervention period
  WBC measures the total number of white blood cells in the blood, reflecting the body's immune response. This is typically measured by collecting a blood sample from venous draw, and analyzed by using an automated blood analyzer.
Blood Routine Test: Red Blood Cell Count (RBC) | From the date of randomization until the end of the 24-week intervention period
  RBC indicates the total number of red blood cells.The measurement involves drawing a blood sample from venous draw and using automated hematological analyzers or manual microscopic methods to count the number of red blood cells.
Blood Routine Test:Hemoglobin | From the date of randomization until the end of the 24-week intervention period
  Hemoglobin is the iron-containing protein in red blood cells that carries oxygen. Its level is measured spectrophotometrically or by hemoglobinometers after collecting a blood sample, providing insights into the blood's oxygen-carrying capacity.
Blood Routine Test:Packed Cell Volume | From the date of randomization until the end of the 24-week intervention period
  Packed Cell Volume measures the percentage of blood volume occupied by red blood cells. It is determined by centrifuging a blood sample to separate the red blood cells from the plasma and measuring the volume occupied by the packed red blood cells.
Blood Routine Test:Platelet Count | From the date of randomization until the end of the 24-week intervention period
  Platelet Count represents the number of platelets in the blood, essential for blood clotting, and low levels can cause bleeding tendencies while high levels may indicate inflammation or other disorders.
Blood Routine Test:Neutrophil Count | From the date of randomization until the end of the 24-week intervention period
  Neutrophil Count reflects the number of neutrophils, a type of white blood cell that plays a key role in fighting bacterial infections, and elevated levels often indicate an active infection or inflammation.
Blood Routine Test:Lymphocyte Count | From the date of randomization until the end of the 24-week intervention period
  Lymphocyte Count measures the number of lymphocytes, another type of white blood cell involved in immune responses, particularly against viral infections, and changes in lymphocyte count can suggest immune system alterations or viral infections.
Urine Routine Test:Urine pH | From the date of randomization until the end of the 24-week intervention period
  Urine pH measures the acidity or alkalinity of urine, crucial for reflecting the body's acid-base balance and the kidney's regulatory function. The normal range is generally between 4.6 and 8.0, with an average of 6.0. This test is conducted using urine analyzers or other methods, and deviations may indicate conditions such as diabetes, gout, acidosis, or frequent vomiting.
Urine Routine Test:Urine Protein | From the date of randomization until the end of the 24-week intervention period
  Urine protein detects the presence of protein in urine, which may indicate kidney disease or other underlying health issues.
Urine Routine Test:Occult Blood | From the date of randomization until the end of the 24-week intervention period
  Occult blood refers to the presence of RBCs in urine that is not visible to the naked eye but can be detected microscopically. This test is usually performed using fresh morning urine, and a positive result may suggest conditions such as urinary tract infections, stones, or kidney diseases.
Urine Routine Test:Red Blood Cells | From the date of randomization until the end of the 24-week intervention period
  Red blood cells in urine are detected through microscopic examination of the urine sediment. More than 3 RBCs per high-power field indicating hematuria. This may be due to kidney bleeding, urinary tract bleeding, or increased glomerular permeability.
Urine Routine Test:White Blood Cells | From the date of randomization until the end of the 24-week intervention period
  White blood cells in urine are also identified via microscopic examination of the urine sediment. Elevated WBCs may indicate infection or inflammation, with normal levels being less than 5 WBCs per HPF.
Urine Routine Test:Urine ketones | From the date of randomization until the end of the 24-week intervention period
  Increased Urine ketones may suggest conditions such as diabetic ketoacidosis, hunger, excessive alcohol consumption, or vigorous exercise.
Renal Function Tests：Creatinine | From the date of randomization until the end of the 24-week intervention period
  Creatinine is a metabolite produced by muscle metabolism and excreted by the kidneys. It serves as an important indicator of renal function.
Renal Function Tests：Estimated Glomerular Filtration Rate (eGFR) | From the date of randomization until the end of the 24-week intervention period
  eGFR is an estimation used to assess kidney function by calculating the rate at which the kidneys filter blood. It is derived from factors including serum creatinine levels, age, gender by using standardized formulas such as MDRD. The measurement provides an indication of renal function and aids in the diagnosis and management of chronic kidney disease. Lower eGFR values indicate decreased kidney function.
Hepatic Function Tests：Aspartate Aminotransferase (AST) | From the date of randomization until the end of the 24-week intervention period
  AST is an enzyme found in multiple tissues, including the liver, heart and skeletal muscle. Elevated AST indicates liver damage.
Hepatic Function Tests：Alanine Aminotransferase (ALT) | From the date of randomization until the end of the 24-week intervention period
  ALT is an enzyme predominantly found in liver cells and is involved in protein metabolism. Elevated ALT indicates liver damage.
Hepatic Function Tests：Glutamyl Transferase (GGT) | From the date of randomization until the end of the 24-week intervention period
  GGT is an enzyme found in the liver and biliary system, and its level is used to detect bile duct issues or liver damage.
QT interval on 18-lead electrocardiogram（ECG） | From the date of randomization until the end of the 24-week intervention period
  The QT interval on 18-lead electrocardiogram（ECG）represents the total duration of ventricular depolarization and repolarization, measured from the beginning of the QRS complex to the end of the T wave.The prolongation of the QT interval may be correlated with drug-induced severe arrhythmias, notably including Torsades de Pointes, thereby making the QT interval one of the key indicators reflecting drug safety.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Hospital of Chengdu University of Traditional Chinese Medicine, Chengdu, Sichuan
  - Deyang Hospital Affiliated to Chengdu University of Traditional Chinese Medicine, Deyang, Sichuan
  - Guangyuan North Sichuan Diabetes Specialty Hospital, Guangyuan, Sichuan

IPD SHARING:
Plan to Share IPD: Yes
Demographic data, including age, gender, and ethnicity of the participants. Baseline clinical data such as blood glucose levels, blood pressure, and diabetes duration.
  Imaging data from multimodaleye - brain imaging, which are anonymized and de - identified to protect patient privacy.
  Outcome data related to the assessment of diabetes neurovascular coupling, like TCM symptom scores and specific functional scores.
  Safety indicators, such as blood and urine routine tests, electrocardiogram
Supporting Information: Study Protocol, CSR
Time Frame: Beginning 1 year after publication and ending 2 years after the publication of results
Access Criteria: The data that support the findings of this study are available from the corresponding author upon reasonable request.

REFERENCES:
- [Background] Mondal R, Deb S, Chowdhury D, Sarkar S, Guha Roy A, Shome G, Sarkar V, Lahiri D, Benito-Leon J. Neurometabolic substrate transport across brain barriers in diabetes mellitus: Implications for cognitive function and neurovascular health. Neurosci Lett. 2024 Nov 20;843:138028. doi: 10.1016/j.neulet.2024.138028. Epub 2024 Oct 24. PMID 39461703
- [Background] Martins B, Pires M, Ambrosio AF, Girao H, Fernandes R. Contribution of extracellular vesicles for the pathogenesis of retinal diseases: shedding light on blood-retinal barrier dysfunction. J Biomed Sci. 2024 May 10;31(1):48. doi: 10.1186/s12929-024-01036-3. PMID 38730462
- [Background] American Diabetes Association Professional Practice Committee. 2. Diagnosis and Classification of Diabetes: Standards of Care in Diabetes-2024. Diabetes Care. 2024 Jan 1;47(Suppl 1):S20-S42. doi: 10.2337/dc24-S002. PMID 38078589